CLINICAL TRIAL: NCT01987479
Title: Multi-Center, Open Label, Single Arm Phase IIIB Study on Safety and Efficacy of Subcutaneous Tocilizumab in Monotherapy or in Combination With Methotrexate or Other Non-Biologic Disease Modifying Antirheumatic Drugs in Rheumatoid Arthritis Patients With an Inadequate Response to Non-Biologic DMARDs - OSCAR
Brief Title: A Study on Safety and Efficacy of Tocilizumab (RoActemra/Actemra) Alone or in Combination With Non-Biologic Antirheumatics in Participants With Rheumatoid Arthritis
Acronym: OSCAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28702; 2013-000342-19 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-19 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tocilizumab Alone or in Combination with Methotrexate or DMARD (Experimental): Participants will receive a weekly SC injection of tocilizumab 162 milligrams (mg) as monotherapy or in combination with methotrexate or other non-biologic DMARDs for 24 weeks.
  Interventions: Drug: Non-Biologic DMARDs; Drug: Tocilizumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Non-Biologic DMARDs — Treatment with non-biologic DMARDs, at a stable dose that was initiated at least 4 weeks prior to baseline, is permitted during the study and is at the investigator's discretion.
Drug: Tocilizumab — Tocilizumab 162 mg will be administered once a week by SC injection and as a single fixed dose, irrespective of body weight, for the treatment duration of 24 weeks.
  Other Names: RoActemra, Actemra
Drug: Methotrexate — Methotrexate will be administered per investigator's discretion.

SUMMARY:
This multi-center, open-label single arm Phase IIIb study will evaluate the safety and efficacy of subcutaneous (SC) tocilizumab administered as monotherapy and/or in combination with methotrexate or other non-biologic disease modifying antirheumatic drugs (DMARDs) in participants with rheumatoid arthritis (RA) with an inadequate response to non-biologic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of active RA according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria.
* Oral corticosteroids (≤10 mg/day prednisone or equivalent), nonsteroidal anti-inflammatory drugs (NSAIDs) and non-biologic DMARDs are permitted if on a stable dose regimen for greater than or equal to (≥]) 4 weeks prior to Baseline.
* Use of effective contraception throughout the study as defined by protocol; female participants of childbearing potential cannot be pregnant.

Exclusion Criteria:

* Presence of clinically significant medical conditions.
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower gastrointestinal disease that might predispose to perforation.
* Current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections.
* Any infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks of Screening or oral antibiotics within 2 weeks of Screening.
* Clinically significant findings on laboratory tests.
* Positive hepatitis B surface antigen or hepatitis C antibody.
* Active tuberculosis requiring treatment within the previous 3 years.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years, or breast cancer diagnosed within the previous 20 years.
* History of alcohol, drug, or chemical abuse within 1 year prior to Screening.
* Neuropathies or other conditions that might interfere with pain evaluation.
* Major surgery (including joint surgery) within 8 weeks prior to Screening or planned major surgery within 6 months following Baseline.
* Rheumatic autoimmune disease other than RA, including systemic lupus erythematosis, mixed connective tissue disorder, scleroderma, polymyositis, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's syndrome). Secondary Sjögren's syndrome with RA is permitted.
* Functional Class IV as defined by the ACR Classification of Functional Status in RA.
* Diagnosis of juvenile idiopathic arthritis or juvenile RA, and/or RA before the age of 16 years.
* Prior history of or current inflammatory joint disease other than RA.
* Exposure to tocilizumab (either intravenous or SC) at any time prior to Baseline.
* Treatment with any investigational agent within 4 weeks (or five half-lives of the investigational drug, whichever is longer) of Screening.
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
* Treatment with IV gamma globulin, plasmapheresis within 6 months of Baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Netherlands (20):
  - ZGT Almelo; Reumatologie, Almelo
  - Jan Van Breemen Instituut, Amsterdam
  - Gelre Ziekenhuizen; Reumatologie, Apeldoorn
  - Amphia ziekenhuis, locatie langendijk, Breda
  - Albert Schweitzer Ziekenhuis ; Dordwijk, Dordrecht
  - Universitair Medisch Centrum Groningen; Department of Rheumatology, Groningen
  - Martini Ziekenhuis, Groningen
  - Kennemer Gasthuis, Haarlem
  - Atrium Medisch Centrum, Heerlen
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - Medisch Centrum Leeuwarden; Reumatology, Leeuwarden
  - Academisch Ziekenhuis Leiden; Dept of Rheumatology, Leiden
  - Maastricht University Medical Centre; Rheumatology, Maastricht
  - Erasmus Medisch Centrum; Reumatologie, Rotterdam
  - Maasstadziekenhuis; Reumatologie, Rotterdam
  - Vlietland Hospital, Schiedam
  - Antonius Ziekenhuis Sneek; Department of Rheumatology, Sneek
  - Leyenburg Ziekenhuis; Internal Medecine, The Hague
  - St. Bronovo-Nebo, The Hague
  - University Medical Centre Utrecht; Reumatologie en Klinische Immunologie, Utrecht

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 174 participants were screened, out of which 150 participants met eligibility criteria and were enrolled into the study.
Groups:
- Tocilizumab Alone or in Combination With Methotrexate or DMARD: Participants received a weekly subcutaneous (SC) injection of tocilizumab 162 milligrams (mg) as monotherapy or in combination with methotrexate or other non-biologic disease modifying antirheumatic drugs (DMARDs) for 24 weeks.
Period: Overall Study
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Started | 150
Completed | 133
Not Completed | 17
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 2
Not completed — Participant/legal guardian decision | 1
Not completed — Other | 5
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all participants who received at least one dose of SC tocilizumab.
Groups:
- Tocilizumab Alone or in Combination With Methotrexate or DMARD: Participants received a weekly SC injection of tocilizumab 162 mg as monotherapy or in combination with methotrexate or other non-biologic DMARDs for 24 weeks.
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.85 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Adverse events included serious as well as non-serious adverse events.
Time Frame: Baseline up to Week 32
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants | 91.3

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR) Score at Weeks 2, 4, 8, 12, 16, 20, 24, and Early Withdrawal
Description: DAS28 was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, erythrocyte sedimentation rate (ESR; millimeters per hour [mm/hour]), and patient's global assessment of disease activity (measured on a 0 to 100 mm Visual Analog Scale [VAS] where 0 mm=no disease activity and 100 mm=worst disease activity). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. Total score range: 0-10, higher score=higher disease activity. DAS28-ESR less than or equal to (≤) 3.2 implied low disease activity and greater than (>) 3.2 to 5.1 implied moderate to high disease activity, and DAS28-ESR less than (<) 2.6 implied clinical remission.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
units on a scale
  Baseline (n=150) | 4.8 (1.3)
  Change at Week 2 (n=148) | 1.337 (0.989)
  Change at Week 4 (n=144) | 2.037 (0.991)
  Change at Week 8 (n=136) | 2.635 (1.098)
  Change at Week 12 (n=133) | 2.908 (1.135)
  Change at Week 16 (n=128) | 3.014 (1.240)
  Change at Week 20 (n=122) | 3.169 (1.170)
  Change at Week 24 (n=121) | 3.232 (1.247)
  Change at early withdrawal visit (n=27) | 1.653 (1.562)

3. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology Criteria 20 (ACR20) Response
Description: A participant had an ACR20 response if there was at least a 20 percent (%) improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either C-reactive protein [CRP] or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2 (n=148) | 20.3 (0.989)
  Week 4 (n=144) | 40.3 (0.991)
  Week 8 (n=136) | 58.1 (1.098)
  Week 12 (n=133) | 69.9 (1.135)
  Week 16 (n=130) | 71.5 (1.240)
  Week 20 (n=123) | 78.9 (1.170)
  Week 24 (n=121) | 82.6 (1.247)
  Early withdrawal visit (n=27) | 37.0 (1.562)

4. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response
Description: A participant had an ACR50 response if there was at least a 50% improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2 (n=148) | 6.1 (0.989)
  Week 4 (n=144) | 18.1 (0.991)
  Week 8 (n=136) | 33.1 (1.098)
  Week 12 (n=133) | 43.6 (1.135)
  Week 16 (n=130) | 52.3 (1.240)
  Week 20 (n=123) | 54.5 (1.170)
  Week 24 (n=121) | 62.0 (1.247)
  Early withdrawal visit (n=27) | 18.5 (1.562)

5. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response
Description: A participant had an ACR70 response if there was at least a 70% improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2 (n=148) | 1.4 (0.989)
  Week 4 (n=144) | 6.9 (0.991)
  Week 8 (n=136) | 14.0 (1.098)
  Week 12 (n=133) | 21.1 (1.135)
  Week 16 (n=130) | 29.2 (1.240)
  Week 20 (n=123) | 38.2 (1.170)
  Week 24 (n=121) | 35.5 (1.247)
  Early withdrawal visit (n=27) | 14.8 (1.562)

6. Secondary Outcome: Percentage of Participants Achieving an ACR90 Response
Description: A participant had an ACR90 response if there was at least a 90% improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2 (n=148) | 0.0 (0.989)
  Week 4 (n=144) | 1.4 (0.991)
  Week 8 (n=136) | 2.9 (1.098)
  Week 12 (n=133) | 6.8 (1.135)
  Week 16 (n=130) | 9.2 (1.240)
  Week 20 (n=123) | 11.4 (1.170)
  Week 24 (n=121) | 15.7 (1.247)
  Early withdrawal visit (n=27) | 3.7 (1.562)

7. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response (Good, Moderate or No Response) Based on DAS28-ESR
Description: DAS28-ESR was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and patient's global assessment of disease activity (VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. The DAS28-ESR based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline >1.2 with a DAS28 score ≤3.2; moderate responders had a change from baseline >1.2 with a DAS28 score >3.2 or a change from baseline >0.6 to ≤1.2 with a DAS28 score ≤5.1. Participants with change from baseline >0.6 to ≤1.2 with a DAS28 score >5.1, or any score with change from baseline ≤0.6, were assessed as non-responders.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2: Good response (n=148) | 34.5 (0.989)
  Week 2: Moderate response (n=148) | 41.9 (0.991)
  Week 2: No response (n=148) | 23.6 (1.098)
  Week 4: Good response (n=144) | 59.7 (1.135)
  Week 4: Moderate response (n=144) | 34.0 (1.240)
  Week 4: No response (n=144) | 6.3 (1.170)
  Week 8: Good response (n=136) | 78.7 (1.247)
  Week 8: Moderate response (n=136) | 17.6 (1.562)
  Week 8: No response (n=136) | 3.7
  Week 12: Good response (n=133) | 85.0
  Week 12: Moderate response (n=133) | 12.0
  Week 12: No response (n=133) | 3.0
  Week 16: Good response (n=128) | 89.1
  Week 16: Moderate response (n=128) | 7.0
  Week 16: No response (n=128) | 3.9
  Week 20: Good response (n=122) | 91.8
  Week 20: Moderate response (n=122) | 5.7
  Week 20: No response (n=122) | 2.5
  Week 24: Good response (n=121) | 92.6
  Week 24: Moderate response (n=121) | 5.0
  Week 24: No response (n=121) | 2.5
  Early withdrawal visit: Good response (n=27) | 44.4
  Early withdrawal visit: Moderate response (n=27) | 29.6
  Early withdrawal visit: No response (n=27) | 25.9

8. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 8, 12, 16, 20, 24, and Early Withdrawal
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, patient and physician global assessment of disease activity assessed on 0-10 centimeter (cm) VAS (0 cm= no disease activity and 10 cm= worst disease activity), and CRP in milligrams per liter (mg/L). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity .
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome. "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 145
units on a scale
  Baseline (n=145) | 26.03 (12.55)
  Change at Week 2 (n=97) | -6.2 (7.4)
  Change at Week 4 (n=78) | -11.3 (8.0)
  Change at Week 8 (n=64) | -14.4 (9.2)
  Change at Week 12 (n=63) | -17.2 (10.8)
  Change at Week 16 (n=67) | -18.5 (11.1)
  Change at Week 20 (n=57) | -19.7 (11.2)
  Change at Week 24 (n=56) | -19.9 (11.8)
  Change at early withdrawal visit (n=18) | -8.0 (10.7)

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 8, 16, 20, 24, and Early Withdrawal
Description: The CDAI is the numerical sum of four outcome parameters: TJC and SJC based on a 28-joint assessment, patient and physician's global assessment of disease activity assessed on 0-10 cm VAS (0 cm= no disease activity and 10 cm= worst disease activity). CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
units on a scale
  Baseline (n=150) | 24.32 (11.84)
  Change at Week 2 (n=148) | -4.7 (7.3)
  Change at Week 4 (n=144) | -9.4 (7.2)
  Change at Week 8 (n=135) | -13.4 (8.7)
  Change at Week 12 (n=132) | -15.4 (9.2)
  Change at Week 16 (n=129) | -16.7 (10.1)
  Change at Week 20 (n=122) | -17.8 (10.2)
  Change at Week 24 (n=121) | -18.3 (11.1)
  Change at early withdrawal visit (n=27) | -6.4 (10.3)

10. Secondary Outcome: Change From Baseline in Total TJC at Weeks 2, 4, 8, 12, 16, 20, 24, and Early Withdrawal
Description: Number of tender joints was determined by examining 28 joints for TJC28 and 68 joints for TJC68, and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28 for a TJC28 and 68 for a TJC68. A reduction in number of tender joints compared to baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
tender joints
  TJC28: Baseline (n=150) | 7.7 (6.5)
  TJC28: Change at Week 2 (n=148) | -1.38 (3.71)
  TJC28: Change at Week 4 (n=144) | -2.94 (3.89)
  TJC28: Change at Week 8 (n=136) | -4.33 (4.82)
  TJC28: Change at Week 12 (n=133) | -4.68 (5.05)
  TJC28: Change at Week 16 (n=130) | -5.36 (5.55)
  TJC28: Change at Week 20 (n=123) | -5.79 (5.24)
  TJC28: Change at Week 24 (n=121) | -5.96 (5.67)
  TJC28: Change at early withdrawal visit (n=27) | -1.07 (4.59)
  TJC68: Baseline (n=150) | 13.2 (10.0)
  TJC68: Change at Week 2 (n=148) | -2.40 (5.84)
  TJC68: Change at Week 4 (n=144) | -5.15 (6.25)
  TJC68: Change at Week 8 (n=136) | -7.19 (7.57)
  TJC68: Change at Week 12 (n=133) | -7.98 (8.46)
  TJC68: Change at Week 16 (n=130) | -9.45 (9.07)
  TJC68: Change at Week 20 (n=123) | -9.86 (9.04)
  TJC68: Change at Week 24 (n=121) | -10.02 (8.94)
  TJC68: Change at early withdrawal visit (n=27) | -1.93 (8.53)

11. Secondary Outcome: Change From Baseline in Total SJC at Weeks 2, 4, 8, 12, 16, 20, 24, and Early Withdrawal
Description: Number of swollen joints was determined by examination of 28 joints for SJC28 and 66 joints for SJC66 and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28 for a SJC28 and 66 for a SJC66. A reduction in number of swollen joints compared to baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and at Early Withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
swollen joints
  SJC28: Baseline (n=150) | 6.2 (5.4)
  SJC28: Change at Week 2 (n=148) | -1.18 (3.04)
  SJC28: Change at Week 4 (n=144) | -2.44 (3.33)
  SJC28: Change at Week 8 (n=136) | -3.62 (3.86)
  SJC28: Change at Week 12 (n=133) | -4.24 (4.17)
  SJC28: Change at Week 16 (n=130) | -4.61 (4.14)
  SJC28: Change at Week 20 (n=123) | -4.92 (4.24)
  SJC28: Change at Week 24 (n=121) | -5.23 (4.63)
  SJC28: Change at early withdrawal visit (n=27) | -1.33 (4.18)
  SJC66: Baseline (n=150) | 9.1 (7.3)
  SJC66: Change at Week 2 (n=148) | -1.84 (4.16)
  SJC66: Change at Week 4 (n=144) | -3.94 (4.35)
  SJC66: Change at Week 8 (n=136) | -5.61 (4.74)
  SJC66: Change at Week 12 (n=133) | -6.50 (5.79)
  SJC66: Change at Week 16 (n=130) | -6.78 (5.95)
  SJC66: Change at Week 20 (n=123) | -7.52 (6.44)
  SJC66: Change at Week 24 (n=121) | -7.80 (6.86)
  SJC66: Change at early withdrawal visit (n=27) | -2.33 (4.89)

12. Secondary Outcome: Percentage of Participants With Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) Dose Reductions or Discontinuation Categorized by Reasons
Description: Results are reported for percentage of participants who had NSAIDs dose reductions or discontinuation by reasons for dose reductions or discontinuation (unknown reasons, safety reasons, other reasons, lack of efficacy, and discomfort).
Time Frame: From Week 16 and before Week 20; From Week 20 and before Week 24
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Unknown reasons (Week 16 to Week 20) | 0.0
  Safety reasons (Week 16 to Week 20) | 0.7
  Other reasons (Week 16 to Week 20) | 0.7
  Lack of efficacy (Week 16 to Week 20) | 0.0
  Discomfort (Week 16 to Week 20) | 0.0
  Unknown reasons (Week 20 to Week 24) | 0.0
  Safety reasons (Week 20 to Week 24) | 0.0
  Other reasons (Week 20 to Week 24) | 0.0
  Lack of efficacy (Week 20 to Week 24) | 0.0
  Discomfort (Week 20 to Week 24) | 0.0

13. Secondary Outcome: Percentage of Participants With Corticosteroid Dose Reductions or Discontinuation Categorized by Reasons
Description: Results are reported for percentage of participants who had corticosteroid dose reductions or discontinuation by reasons for dose reductions or discontinuation (unknown reasons, safety reasons, other reasons, lack of efficacy, and discomfort).
Time Frame: From Week 16 and before Week 20; From Week 20 and before Week 24
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Unknown reasons (Week 16 to Week 20) | 0.0
  Safety reasons (Week 16 to Week 20) | 1.3
  Other reasons (Week 16 to Week 20) | 0.7
  Lack of efficacy (Week 16 to Week 20) | 0.0
  Discomfort (Week 16 to Week 20) | 0.0
  Unknown reasons (Week 20 to Week 24) | 0.0
  Safety reasons (Week 20 to Week 24) | 0.0
  Other reasons (Week 20 to Week 24) | 1.3
  Lack of efficacy (Week 20 to Week 24) | 0.7
  Discomfort (Week 20 to Week 24) | 0.0

14. Secondary Outcome: Time to Discontinuation or First Dose Reduction of Corticosteroids or NSAIDs
Description: Time to discontinuation or first dose reduction of corticosteroids or NSAIDs (weeks) = (Date of the first dose reduction or end date of corticosteroids or NSAIDs treatment - date of first drug intake of this study) + 1. Time to discontinuation or first dose reduction was based on the first occurring event (corticosteroid discontinuation or corticosteroid first dose reduction or NSAIDs discontinuation or NSAIDs first dose reduction, whichever occurred first).
Time Frame: Baseline up to Week 32
Population: FAS population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
weeks | 25.3 [25.0 to 28.0]

15. Secondary Outcome: Percentage of Participants With Anti-Tocilizumab Antibodies
Time Frame: Baseline, Weeks 12 and 24, early withdrawal (up to Week 24), follow-up visit (8 weeks after last dose of tocilizumab, up to 32 weeks)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Baseline (n=147) | 6.1 (0.5906)
  Week 12 (n=5) | 40.0 (0.5734)
  Week 24 (n=121) | 7.4 (0.5587)
  Early withdrawal (n=22) | 9.1 (0.5330)
  Follow-up visit (n=26) | 11.5 (0.5682)

16. Secondary Outcome: Serum Levels of Tocilizumab
Time Frame: as for outcome 15
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
micrograms per milliliter (mcg/mL)
  Baseline (n=4) | 0.5 (0.3)
  Week 12 (n=123) | 42.3 (25.2)
  Week 24 (n=112) | 46.5 (29.2)
  Early withdrawal (n=17) | 16.8 (19.3)
  Follow-up visit (n=3) | 60.9 (29.7)

17. Secondary Outcome: Serum Levels of Soluble Interleukin-6 Receptors (sIL-6Rs)
Time Frame: as for outcome 15
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
nanograms per milliliter (ng/mL)
  Baseline (n=139) | 38.3 (10.4)
  Week 12 (n=126) | 516.6 (137.7)
  Week 24 (n=115) | 536.5 (161.6)
  Early withdrawal (n=21) | 380.4 (215.2)
  Follow-up visit (n=26) | 117.5 (194.3)

18. Secondary Outcome: Patient Global Assessment of Disease Activity VAS Scores
Description: Patient global assessment of disease activity was measured on a 0 to 100 mm horizontal VAS where 0 mm=no disease activity and 100 mm=maximum disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and Early withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
mm
  Baseline (n=150) | 54.8 (22.3)
  Week 2 (n=148) | 43.6 (23.0)
  Week 4 (n=144) | 35.5 (23.0)
  Week 8 (n=136) | 27.2 (21.8)
  Week 12 (n=133) | 22.2 (20.3)
  Week 16 (n=129) | 21.3 (21.0)
  Week 20 (n=123) | 19.2 (18.6)
  Week 24 (n=121) | 18.8 (19.5)
  Early withdrawal (n=27) | 40.4 (30.9)

19. Secondary Outcome: Patient Pain VAS Scores
Description: This assessment represents the participant's assessment of his/her current level of pain on a 100 mm horizontal VAS where 0 mm= no pain to 100 mm= unbearable pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and Early withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
mm
  Baseline (n=150) | 52.5 (22.1)
  Week 2 (n=148) | 44.4 (21.9)
  Week 4 (n=144) | 35.8 (22.3)
  Week 8 (n=136) | 27.6 (21.3)
  Week 12 (n=133) | 21.7 (19.0)
  Week 16 (n=129) | 20.9 (20.2)
  Week 20 (n=123) | 19.5 (18.0)
  Week 24 (n=121) | 19.6 (18.8)
  Early withdrawal (n=27) | 42.8 (30.4)

20. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire measures functional status (disability) and health-related quality of life. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question is evaluated according to the degree of severity on a 4-point scale. Total score for HAQ-DI was the average of all questions and ranges from 0 = without any difficulty to 3 = unable to do.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and early withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
units on a scale
  Baseline (n=147) | 1.2329 (0.5708)
  Week 2 (n=147) | 1.0978 (0.5906)
  Week 4 (n=143) | 0.9673 (0.5734)
  Week 8 (n=134) | 0.8249 (0.5587)
  Week 12 (n=131) | 0.7460 (0.5330)
  Week 16 (n=129) | 0.6996 (0.5682)
  Week 20 (n=122) | 0.6620 (0.5333)
  Week 24 (n=119) | 0.6681 (0.5745)
  Early withdrawal (n=27) | 1.2315 (0.6853)

21. Secondary Outcome: Percentage of Participants Compliant to Tocilizumab Treatment as Measured by Diary Cards and Return Records
Description: A diary card was provided to participants to record home injections. Participants were asked to return all empty drug supply boxes, unused pre-filled syringe, and diary cards to the clinic at each visit as a measure of drug accountability and participant compliance. A participant was considered compliant if the participant correctly administered all scheduled doses of SC tocilizumab during the assessment period.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, and early withdrawal (up to Week 24)
Population: FAS population. "n" = participants who were evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
percentage of participants
  Week 2 (n=148) | 90.5 (0.5906)
  Week 4 (n=144) | 95.8 (0.5734)
  Week 8 (n=136) | 91.9 (0.5587)
  Week 12 (n=133) | 97.7 (0.5330)
  Week 16 (n=130) | 93.8 (0.5682)
  Week 20 (n=123) | 95.1 (0.5333)
  Week 24 (n=121) | 92.6 (0.5745)
  Early withdrawal (n=27) | 88.9 (0.6853)

22. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: The FACIT-F score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, and early withdrawal (up to Week 24)
Population: FAS population. Here, "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Number analyzed (Participants) | 150
units on a scale
  Baseline (n=133) | 29.84 (9.43)
  Week 2 (n=134) | 33.07 (9.34)
  Week 4 (n=133) | 35.10 (10.37)
  Week 8 (n=126) | 37.34 (9.25)
  Week 12 (n=126) | 37.89 (8.52)
  Week 16 (n=122) | 37.93 (9.11)
  Week 20 (n=118) | 39.65 (8.87)
  Week 24 (n=114) | 39.93 (8.65)
  Early withdrawal (n=27) | 33.48 (12.06)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 32
Description: FAS population
Arm/Group | Tocilizumab Alone or in Combination With Methotrexate or DMARD
Serious Adverse Events (participants affected / at risk) | 14/150
Other Adverse Events (participants affected / at risk) | 77/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Alone or in Combination With Methotrexate or DMARD (N=150)
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Prophylaxis (Surgical and medical procedures) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Alone or in Combination With Methotrexate or DMARD (N=150)
Nasopharyngitis (Infections and infestations) | 35
Nausea (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 18
Dizziness (Nervous system disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.